CLINICAL TRIAL: NCT00559702
Title: A Randomized, Open-Label, Dose-Ranging Study to Evaluate the Pharmacokinetics and Initial Safety of Subcutaneous and Intramuscular Natalizumab in Subjects With Multiple Sclerosis
Brief Title: Safety Study of Natalizumab to Treat Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101MS102
Record Dates: First submitted 2007-11-07; First posted 2007-11-16 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
Keywords: natalizumab; multiple sclerosis; Tysabri ®
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Natalizumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Natalizumab IV (Participants with secondary progressive multiple sclerosis)
  Interventions: Drug: natalizumab
- 2 (Experimental): Natalizumab IM (Participants with secondary progressive multiple sclerosis)
  Interventions: Drug: natalizumab
- 3 (Experimental): Natalizumab SC (Participants with secondary progressive multiple sclerosis)
  Interventions: Drug: natalizumab
- 4 (Other): Standard of care as determined by the Investigator and Treating Neurologist (Participants with secondary progressive multiple sclerosis)
  Interventions: Other: standard of care
- 5 (Experimental): Natalizumab SC (Participants with relapsing forms of multiple sclerosis)
  Interventions: Drug: natalizumab
- 6 (Experimental): Natalizumab IV (Participants with relapsing forms of multiple sclerosis)
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab — natalizumab
  Other Names: Tysabri ®; BG00002
  Arms: 1; 2; 3; 5; 6
Other: standard of care — standard of care as determined by the Investigator and Treating Neurologist
  Arms: 4

SUMMARY:
The primary objective of this study is to compare the pharmacokinetic (PK) and pharmacodynamics (PD) of single subcutaneous (SC) and intramuscular (IM) doses of 300 mg natalizumab to intravenous (IV) administration of 300 mg natalizumab in multiple sclerosis (MS) participants. The secondary objectives are to investigate the safety, tolerability and PK of repeated natalizumab doses administered SC and IM, to investigate the immunogenicity of repeated natalizumab doses administered SC and IM, to explore proof of concept within the secondary progressive multiple sclerosis (SPMS) population using change from baseline in clinical measures including: expanded disability status scale (EDSS), multiple sclerosis functional composite scale (MSFC), symbol digit modalities test (SDMT), visual analogue scale (VAS), and visual function test; and brain magnetic resonance imaging (MRI) measures including: number of new or newly-enlarging T2 hyperintense lesions, number of new T1 hypointense lesions, number of new gadolinium-enhancing (Gd+) lesions, whole brain atrophy, magnetization transfer ratio (MTR), and diffusion tensor imaging (DTI) and to observe the effect of natalizumab administered IV and SC on brain MRI measures in participants with relapsing forms of MS.

ELIGIBILITY:
Key Inclusion Criteria:

* For arms 1,2,3 and 4: Diagnosis of Secondary Progressive Multiple Sclerosis (SPMS)
* For arms 5 and 6: Diagnosis of relapsing forms of Multiple Sclerosis (MS).
* No past history of receiving natalizumab.

Key Exclusion Criteria:

* For arms 1,2,3 and 4 Diagnosis of primary progressive MS or relapsing-remitting MS.
* Form arms 5 and 6: Diagnosis of primary progressive MS or secondary progressive MS without the occurrence of relapses.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of natalizumab | Pre-dose, 4, 24, 48, 72 and 96 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
Time to maximum observed concentration (Tmax) of natalizumab | Pre-dose, 4, 24, 48, 72 and 96 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
Area under the curve to the last measurable concentration (AUC0-last) of natalizumab | Pre-dose, 4, 24, 48, 72 and 96 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
  Area under the curve to the last measurable concentration as measured by the trapezoidal rule.
Apparent volume of distribution of natalizumab | Pre-dose, 4, 24, 48, 72 and 96 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
Half-life of natalizumab | Pre-dose, 4, 24, 48, 72 and 96 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
Area under the curve extrapolated to infinity (AUC0-∞) of natalizumab | Pre-dose, 4, 24, 48, 72 and 96 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
Apparent Clearance of natalizumab | Pre-dose, 4, 24, 48, 72 and 96 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
α4-integrin saturation | Pre-dose, 4, 24 and 72 hours post-dose and Days 7, 14, 21, 28, 35, 42 and 56
  PD activity will be assessed by measuring the degree of natalizumab saturation of the very late antigen-4 (also known as α4β1 integrin) VLA-4 (α4β1) receptor on peripheral blood lymphocyte/monocyte populations.

SECONDARY OUTCOMES:
Number of Participants with adverse events | 13-19 months
Number of participants with abnormalities in vital signs | 13-19 months
Number of participants with changes in the physical examination | 13-19 months
Number of participants with abnormal laboratory test results | 13-19 months
Number of participants with natalizumab antibodies | Days 28, 42, 56, Weeks 24 and 32
Change from Baseline in expanded disability status scale (EDSS) | Baseline, Weeks 8, 20, and 32
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Change form Baseline in Multiple Sclerosis Functional Composite Scale (MFSC) | Baseline, Weeks 8, 20, and 32
  The MFSC consists of 3 tests: 1. Timed 25-Foot Walk, a quantitative mobility and leg function performance test where the participant is timed while walking for 25 feet; 2. 9-Hole Peg Test (9HPT), a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs. 3. 3 Second Paced Auditory Serial Addition Test (PASAT 3). The MSFC is based on the concept that scores for these 3 dimensions - arm, leg, and cognitive function are combined to create a single score that can be used to detect change over time. A composite z-score is created, which represents the number of standard deviations (SDs) a participant's test result is higher (z > 0) or lower (z < 0) than the average test result (z = 0) of the reference population.
Change from Baseline in Symbol Digit Modalities Test (SDMT) | Baseline, Weeks 8, 20, and 32
  SDMT is a screening test for cognitive impairment. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 to 110 (best).
Change from Baseline in visual analog scale (VAS) | Baseline, Weeks 8, 20, and 32
  The participant's global assessment of well-being as assessed using a visual analogue scale (VAS) is a quality of life measurement that will be evaluated for the specified time periods. Participants report how they feel on a scale of 0 to 100, where 0 indicates being "poor" and 100 being "excellent."
Change from Baseline in visual function test | Baseline, Weeks 8, 20, and 32
Number of new or newly enlarging T2 hyperintense lesions | Baseline and Week 32
  Measured by magnetic resonance imaging (MRI).
Number of new gadolinium-enhanced lesions | Baseline and Week 32
  Measured by magnetic resonance imaging (MRI).
Number of new T1 hypointense lesions | Baseline and Week 32
  Measured by magnetic resonance imaging (MRI).
Whole brain atrophy | Baseline and Week 32
  Atrophy will be measured as the percent brain volume change (PBVC) and will be assessed using the Structural Image Evaluation of Normalized Atrophy (SIENA).
Percent change in magnetization transfer ratio (MTR) | Baseline and Week 32
  Remyelination will be measured using magnetization transfer ratio (MTR) in whole brain (WB) and normal-appearing brain tissue (NABT),
Diffusion tensor imaging (DTI) | Baseline and Week 32
Injection site pain assessment | Pre-dose, 5 and 15 minutes and 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- United States (12):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Berkeley, California
  - Research Site, Centennial, Colorado
  - Research Site, Maitland, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Peoria, Illinois
  - Research Site, Farmington Hills, Michigan
  - Research Site, Buffalo, New York
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Vienna, Virginia